CLINICAL TRIAL: NCT05722002
Title: Comparing Analgesic Regimen Effectiveness and Safety for Surgery (CARES) Trial
Acronym: CARES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Mark Bicket, MD, PhD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00215416; CER-2021C1-22398 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-02

CONDITIONS: Surgery; Pain, Postoperative
Keywords: Medications after surgery; NSAIDS; Acetaminophen; Opioids; laparoscopic gallbladder removal; inguinal hernia repair; breast lumpectomy; Analgesics, non-narcotic
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Opioid; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomization of patients will be stratified by site, sex, age (greater or equal to 65 years old), and type of surgery, via permuted block randomization with a variable block size.
Who Masked: Outcomes Assessor
Masking Description: Both study staff performing outcome assessment and data analysis will be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAID regimen (Other): Surgical teams will elect for one of the medications within the treatment arm to which the patient is randomized.
  Interventions: Drug: NSAID; Drug: Acetaminophen
- Opioid regimen (Other)
  Interventions: Drug: Opioid; Drug: Acetaminophen

INTERVENTIONS:
Drug: NSAID — Once randomized to this group the surgical team will elect for 1 of the following treatment options to be given:
  * Ibuprofen 600 milligram (mg) by mouth every six hours as needed for pain (10 doses)
  * Celecoxib 400 mg by mouth once then 200 mg every twelve hours as needed for pain (10 doses)
  * Naproxen 500 mg by mouth once then 250 mg by mouth every eight hours as needed for pain (10 doses)
  Arms: NSAID regimen
Drug: Opioid — Once randomized to this group the surgical team will elect for 1 of the following treatment options to be given:
  * Oxycodone 5 mg by mouth every four to six hours as needed for pain, 10 doses
  * Morphine 7.5 mg by mouth every four to six hours as needed for pain, 10 doses
  * Hydromorphone 2 mg by mouth every four to six hours as needed for pain, 10 doses
  Arms: Opioid regimen
Drug: Acetaminophen — Acetaminophen 1000 mg by mouth every 6 hours around the clock for the first three days after surgery then as needed thereafter (20 doses).

SUMMARY:
This trial is being completed to compare two commonly used options to treat pain after surgery. Participants that undergo gallbladder removal, hernia repair, and breast lump removal will be eligible to enroll. Eligible participants will be randomized to 1 of 2 groups of medications (Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) plus acetaminophen or low dose opioids plus acetaminophen).

It is anticipated that the NSAID group will have superior clinical outcomes and fewer side effects when compared to the opioid group.

ELIGIBILITY:
Inclusion Criteria:

* No significant analgesic medication use before surgery: For this study, significant analgesic medication use before surgery as use of prescriptions for opioid or NSAID medications in the past 30 days, or over-the-counter NSAID use on greater than 7 of 30 past days, as reported by the patient.
* One of three common low-risk surgical procedures: For this study, the three-common low-risk surgical procedures will include laparoscopic gallbladder removal, inguinal hernia repair, and breast lumpectomy.

Exclusion Criteria:

* Anticipated other surgery within 6 months or anticipated life expectancy of less than 6 months
* Patients with contraindications to NSAID drugs in the NSAID arm, opioid drugs in the OPIOID arm, or acetaminophen will be excluded. There are specific contraindications that will be reviewed per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity based on Brief Pain Inventory (BPI) pain intensity score at the surgical site over 7 days post surgery | 7 days post surgery
  This is a one question survey in which the worst pain intensity recorded (0-10 being the worst) will be used.
Safety outcome - number and severity of any adverse medication-related symptoms over 7 days post surgery | 7 days post surgery
  Symptom Checklist will proactively screen patients for reports of adverse events from analgesic medications over the first 7 days post surgery.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance v1.0 4a questionnaire | 1 month post surgery
  This is a 4 question survey in which participants will rate statements pertaining to quality of sleep.
  Participants will also rate sleep quality as very poor (5), poor (4), fair (3), good (2), or very good (1).
Clinically important adverse events | 180 days post surgery
  The study team will review charts for unplanned postoperative clinical interactions related to pain (patient messages, phone calls, non-routine clinic visits related to pain) and emergency room visits, hospitalizations, and 30-day complications after discharge measured using the American College of Surgeons' (ACS) National Surgical Quality Improvement Program (NSQIP) definitions.
Patient Global Impression of Change (PGIC) | up to 1 month after surgery
  The perception of improvement after treatment will be assessed by the patient global impression of change PGIC (range 0-7).
Quality of Recovery (QoR) 15 | 3 days post surgery
  There are 15 questions assessed on a scale of 1-10, with 0 being none of the time and 10 being all of the time, 10 being the better outcome.
Quality of Recovery (QoR) 15 | 7 days post surgery
  There are 15 questions assessed on a scale of 1-10, with 0 being none of the time and 10 being all of the time, 10 being the better outcome.
PROMIS Pain Interference 4a | 3 months
  This is a 4 question survey that assesses the degree to which pain interferes with various aspects of life. Items are scored on a 1 ("Not at all") to 5 ("Very much") scale with a range of 4 - 20. Higher scores indicate greater pain interference.
PROMIS Preference score 29+2 Profile v2.1 | 3 months
  This is a 31 question survey that includes questions to evaluate each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social functioning, and pain interference) using a 5- point Likert scale, as well as a single item to assess pain severity on a 0-10 scale as well as 2 questions for cognitive function. Higher scores are indicative of better health.
Substance use based on the Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) tool | 180 days post surgery
  This National Institute on Drug Abuse (NIDA) TAPS tool has part 1 (5 questions) and part 2 (possible 9 questions).
National Survey on Drug Use and Health Questions (NSDUH) on Opioid Misuse opioid misuse question | 3 months
National Survey on Drug Use and Health Questions (NSDUH) on Opioid Misuse opioid misuse question | 180 days
New prolonged opioid use | days 4-180 post surgery
  This will include greater or equal to 1 opioid prescription post-discharge between 4-180 days post discharge.
Chronic pain based on Brief Pain Inventory (BPI) pain intensity score at 180 days post surgery | 180 days post surgery
  One question survey in which the participants rate pain intensity recorded (0-10), ten being the worst.
Chronic pain based on Body Map | 180 days post surgery
  Participants will document/mark on this image map to identify areas in which persistent or recurrent pain was felt.
Acute pain based on The Michigan Body Map | 7 days post surgery
  Participants will document/mark on this image map to identify areas in which persistent or recurrent pain was felt.
Healthcare Utilization related to pain at 1 month | within 1 months after surgery
  Participants will answer questions about their healthcare utilization related to pain for the time period from date of surgery to one month later for the following three events: (1) postoperative clinical interactions related to pain in the form of patient messages, phone calls, and non-routine clinic visits related to pain, (2) emergency room visits, and (3) hospitalizations. The study team will also review health record for the same events.
Healthcare Utilization related to pain at 6 months | within 6 months after surgery
  Participants will answer questions about their healthcare utilization related to pain for the time period from date of surgery to six months later related to pain for the following three events: (1) postoperative clinical interactions in the form of patient messages, phone calls, and non-routine clinic visits related to pain, (2) emergency room visits, and (3) hospitalizations. The study team will also review health record for the same events.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bicket, MD, PhD, Principal Investigator — University of Michigan
Locations (8):
- United States (6):
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University in Saint Louis, St Louis, Missouri
  - Cooper University Health Care, Camden, New Jersey
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Temple University - Temple Health, Philadelphia, Pennsylvania
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the trial that is not subject to restrictions based on data sharing agreements (e.g., prescription drug monitoring program data), after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anticipated summer of 2028 with no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by a review committee and the sponsor. The type of analyses will be for analyses related to aims in the proposal. Proposals may be submitted up to 36 months after data availability, after which data will be available in the data warehouse but without investigator support.

REFERENCES:
- [Derived] Bicket MC, Ladha KS, Haroutounian S, McFarlin K, Neff M, McDuffie RL, Waljee JF, Wijeysundera DN, Brummet C, Li Y; CARES Investigators. Comparing Analgesic Regimen Effectiveness and Safety after Surgery (CARES): protocol for a pragmatic, international multicentre randomised trial. BMJ Open. 2025 Apr 5;15(4):e099925. doi: 10.1136/bmjopen-2025-099925. PMID 40187774